CLINICAL TRIAL: NCT07235865
Title: Non-Invasive Diagnosis and Monitoring of Cardiac Masses by Liquid Biopsy: The CarMA Study
Brief Title: Non-Invasive Diagnosis and Monitoring of Cardiac Masses by Liquid Biopsy
Acronym: CarMA
Status: Recruiting | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 4861
Record Dates: First submitted 2025-08-23; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Masses
Keywords: Early-Onset Colorectal Cancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- benign cardiac lesions: patients diagnosed with benign cardiac lesions
  Interventions: Genetic: NGS-guided regimen: Regimen A
- primary cardiac sarcomas: patients diagnosed with primary cardiac sarcomas (PCS)
  Interventions: Genetic: NGS-guided regimen: Regimen A

INTERVENTIONS:
Genetic: NGS-guided regimen: Regimen A — Liquid biopsy, consisting of a venous blood sample, will be collected during routine venipuncture
  Other Names: collection of blood for NGS and archival tissue sample, where available

SUMMARY:
This is a nonprofit, observational, prospective and retrospective,multicenter study in a population of young and adult patients ≥12 years with a diagnosis of a cardiac mass. The study will include both patients with masses of unknown pathological diagnosis and patients with a known histology of benign or malignant tumors. We predict a case-control allocation ratio of 1:1 between cardiac malignant tumors and benign lesions. Peripheral blood will be collected at participating centers during routine venipuncture,processed and then shipped for liquid biopsy ctDNA NGS analyses. If available, in malignant cases, matched tumor tissue samples collected as per clinical practice solid biopsies or surgery will be used for analyses. Longitudinal tracking through serial blood draws could be performed in selected cases of patients with cardiac malignancies who receive cancer treatment

DETAILED DESCRIPTION:
This is a nonprofit, observational, prospective and retrospective, multicenter study. The primary objectives of this study are: (i) to assess the efficacy of liquid biopsy using ctDNA NGS in identifying tumor-specific somatic alterations in patients with cardiac malignancies, particularly primary cardiac sarcomas (PCS), and to differentiate these from benign cardiac lesions. Liquid biopsy, consisting of a venous blood samplecollected during routine venipuncture, will assess the nature of circulating DNA by a commercial NGS assay (i.e., Guardant Infinity, Guardant Health) and/or academic assays. When solid biopsy is available since previouslyperformed as per clinical practice, tumor DNA will be assessed by a commercial issue NGS assay (i.e., FoundationOne, Foundation Medicine) and/or academic assays

ELIGIBILITY:
Inclusion Criteria

1. Age ≥12 years old
2. Suspected or confirmed diagnosis of a cardiac mass of any nature as assessed by standard clinical, radiological and/or pathological procedures.

Exclusion Criteria

1. Inability of the pa ent to fully understand and sign the informed consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: control:benign cardiac lesions; case:primary cardiac sarcomas young and adult patients with a diagnosis of a cardiac mass
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Molecular profile | Jul2024-Jul2029
  Collect and analyse blood and tissue samples from both cases and control in terms of molecular profile

SECONDARY OUTCOMES:
Molecular targets | Jul2024-Jul2029
  Collection and alalysis of blood and tissue samples from both cases and control in term of molecular profile.
  To identify the percentage and types of actionable molecular targets that could be amenable of potential targeted treatment according to the ESMO Scale for Clinical Actionability of molecular Targets (ESCAT). To test the concordance of liquid biopsy NGS ctDNA with tissue-based NGS analyses in a subset of patients where both tissue and blood samples are available.

CONTACTS AND LOCATIONS:
Overall Officials: Katia Bencardino, MD, Principal Investigator — Niguarda Hospital
Locations (1):
- Niguarda Hospital, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet